CLINICAL TRIAL: NCT02877069
Title: A Prospective, Single-arm Study of the Safety and Effectiveness of VYC-12 Hyaluronic Acid Injectable Gel for Treatment of Superficial Cutaneous Depressions Such as Fine Lines and for Improvement of Skin Quality
Brief Title: Safety and Effectiveness of VYC-12 Hyaluronic Acid Injectable Gel for Treatment of Superficial Cutaneous Depressions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V12-001
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Skin Roughness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VYC-12 Injectable Gel (Experimental): VYC-12 Hyaluronic Acid (HA) injectable gel administered as an intradermal injection on Day 0 in the face and if applicable neck areas. Participants are eligible to receive up to 3 treatments including an optional top-up and an optional second treatment.
  Interventions: Device: VYC-12 HA injectable gel

INTERVENTIONS:
Device: VYC-12 HA injectable gel — VYC-12 Hyaluronic Acid (HA) injectable gel administered as an intradermal injection.

SUMMARY:
This study will evaluate the safety and effectiveness of VYC-12 hyaluronic acid (HA) injectable gel for filling fine lines, as measured by skin texture improvement, and for improvement of skin quality.

ELIGIBILITY:
Inclusion Criteria:

* Participants in good general health
* Score of 2=Moderate (coarse and uneven visual skin texture) or 3=Severe (coarse visual skin texture, crosshatched fine lines) on both cheeks using the 5-Point Allergan Skin Roughness Scale (ASRS).

Exclusion Criteria:

* Has undergone tissue augmentation with dermal fillers including HA, calcium hydroxylapatite, autologous fat, mesotherapy, or other cosmetic procedures (eg. face-lift, laser, photomodulation, intense pulsed light, radiofrequency, dermabrasion, chemical peel, or other ablative procedures) in the face or neck within the past 12 months
* Has received any crosslinked HA filler in any anatomic area within the past 12 months
* Has undergone treatment with botulinum toxins in the face or neck within the past 6 months
* Has ever received semi-permanent fillers or permanent facial implants (eg. poly-L-lactic acid, polymethylmethacrylate, silicone, expanded polytetrafluoroethylene) anywhere in the face or neck
* Has facial hair that would interfere with the visualization of the face or neck
* Has undergone a dental procedure within the past 6 weeks
* Has a tendency to develop hypertrophic scarring
* Has a history of allergy to HA products and/or to gram-positive bacterial proteins as HA is produced by Streptococcus-type bacteria
* Has a history of anaphylactic shock
* Has been previously diagnosed with streptococcal disease (eg. recurrent sore throat, acute rheumatic fever)
* Has current cutaneous inflammatory or infectious processes (eg. acne, herpes), abscess, an unhealed wound, or a cancerous or precancerous lesion on the face or neck
* Is on an ongoing regimen of anticoagulation therapy (eg. warfarin)
* Is on an ongoing regimen of medications (eg. aspirin, ibuprofen) or other substances (eg, herbal supplements with garlic, gingko biloba, or ginseng) known to increase coagulation time within 10 days of undergoing study device injection
* Has begun using any over-the-counter or prescription, oral or topical, antiwrinkle products on the face or neck within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with a ≥1 Point Improvement in the 5-Point Allergan Skin Roughness Scale (ASRS) compared to Baseline | Baseline, Month 1

SECONDARY OUTCOMES:
Change from Baseline in Instrument Measures of Cheek Skin Smoothness | Baseline, Month 1
Change from Baseline in Instrument Measures of Cheek Skin Hydration | Baseline, Month 1
Change from Baseline in Instrument Measures of Cheek Skin Elasticity | Baseline, Month 1

CONTACTS AND LOCATIONS:
Overall Officials: Nikki Amaratunge, Study Director — Allergan
Locations (1):
- Laboratoire Dermscan-Pharmascan, Lyon, Auvergne-Rhône-Alpes, France

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com